CLINICAL TRIAL: NCT06710561
Title: The Phase I Single-center, Single-blind, Randomized Clinical Study of the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Injectable SPN01
Brief Title: The Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of Injectable SPN01 in Phase I.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing SonoPhotoNano Medical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPN01-Ⅰ-01
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Healthy subjects will receive intravenous injection of different doses of injectable SPN01 and placebo in a single dose.
  Interventions: Drug: SPN01 for Injection; Other: Placebo
- Phase 2 (Experimental): Colorectal cancer subjects will receive intravenous injection of SPN01 0.06 mg/kg for a single dose.
  Interventions: Drug: SPN01 for Injection

INTERVENTIONS:
Drug: SPN01 for Injection — After each subject was randomly assigned, different doses of SPN01 for Injection (0.02 mg/kg, 0.06 mg/kg, 0.12 mg/kg) were administered intravenously in a single dose.
  Arms: Phase 1
Other: Placebo — After each subject was randomly assigned, a single intravenous injection of 0.9% sodium chloride was administered
  Arms: Phase 1
Drug: SPN01 for Injection — Colorectal cancer subjects will receive intravenous injection of SPN01 0.06 mg/kg for a single dose.
  Arms: Phase 2

SUMMARY:
The primary objective of this study is: to evaluate the safety and tolerability of injectable SPN01 in subjects. The secondary objective of this study is: to evaluate the pharmacokinetic characteristics of injectable SPN01 in subjects.The exploratory objectives of this study are: (1)to evaluate the preliminary efficacy of injectable SPN01 in subjects with colorectal cancer. (2) to evaluate the effect of the blood concentration of injectable SPN01 on the QTc interval. (3) to evaluate the metabolic characteristics of injectable SPN01 in humans.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI): BMI between 19.0 kg/m² and 26.0 kg/m² (inclusive). For male subjects, body weight must be ≥50.0 kg; for female subjects, body weight must be ≥45.0 kg.
2. Contraceptive Use: Males or females of childbearing potential must use effective contraception during the study and for 30 days after administration. Effective contraception includes sterilization, intrauterine hormonal devices, condoms, contraceptive pills/devices, abstinence, or vasectomy.
3. Informed Consent: The subject must fully understand the purpose, nature, methods, and potential adverse effects of the study, voluntarily agree to participate, sign a written informed consent form, and comply with the study protocol.
4. For healthy subjects-Age between 18 and 45 years (inclusive), either male or female.
5. For healthy subjects-eGFR ≥ 90 ml/min/1.73 m².
6. For healthy subjects-Screening phase laboratory results (blood count, blood biochemistry, urine routine, coagulation function) must be normal or clinically insignificant.
7. For healthy subjects-Good general health with no major diseases, as determined by the investigator through history, vital signs, physical examination, clinical ECG, and laboratory test results.
8. For colorectal cancer subjects-Age between 18 and 75 years (inclusive), either male or female.
9. For colorectal cancer subjects-Pathologically confirmed diagnosis of colorectal cancer and scheduled for surgery (laparoscopic or open surgery).
10. For colorectal cancer subjects-No prior targeted treatment for colorectal cancer (including radiotherapy, chemotherapy, targeted therapy, etc.).
11. For colorectal cancer subjects-At least one evaluable lesion.

Exclusion Criteria:

1. Pregnancy or Lactation: Female subjects who are pregnant (positive pregnancy test at screening) or breastfeeding.
2. Pregnancy or Donation Plans: Subjects planning to become pregnant or donate sperm/eggs during the study or within 3 months after administration.
3. Allergy to SPN01: Known allergy to any component of the investigational drug SPN01, or a history of severe allergies.
4. History of Severe Systemic Diseases: A history of serious systemic diseases (including cardiovascular, digestive, urinary, respiratory, endocrine, immune, hematological, lymphatic, musculoskeletal, neurological diseases), liver or kidney dysfunction, or psychiatric disorders.
5. Alcohol or Drug Abuse: A history of alcohol or drug abuse/dependence.
6. Severe or Uncontrolled Psychiatric Disorder: Subjects with severe or uncontrolled psychiatric diseases.
7. Active Infection: Any active infection requiring systemic treatment or uncontrolled infection within 14 days prior to the start of the study drug.
8. Infectious Disease Positive: Subjects who test positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or syphilis; subjects who test positive for hepatitis B virus (HBV) surface antigen.
9. Needle Phobia: Subjects with a history of vasovagal response to blood draws or injections and those who cannot tolerate intravenous cannulation.
10. Blood Donation or Blood Loss: Subjects who have donated blood or experienced total blood loss of ≥400 mL within the last 3 months.
11. Medication Use: Subjects who have taken any prescription drugs, over-the-counter medications, or herbal products within 2 weeks prior to the first dose, especially those who have used antacids (e.g., proton pump inhibitors, H2 receptor antagonists), P-glycoprotein (P-gp) inhibitors, or drugs associated with a risk of torsades de pointes, or those who have used any medications within 30 days prior to the first dose that inhibit or induce liver drug metabolism.
12. Other Clinical Trials: Participation in another clinical trial and use of other investigational drugs within 30 days prior to screening.
13. Vaccination: Receipt of any vaccination within 3 months prior to screening or plans to receive a vaccine during the study.
14. Other Conditions: Any other condition that, in the opinion of the investigator, would make the subject unsuitable for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-17 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Predose and up to 24 hours postdose
  Safety and tolerability will be assessed through the monitoring of adverse events (AEs), clinical laboratory tests (including complete blood count, blood biochemistry, coagulation function, and urinalysis), local safety assessments, vital sign checks (including temperature, respiration rate, pulse rate, and blood pressure), 12-lead electrocardiogram (ECG), and physical examinations.
  Adverse events (AEs) and serious adverse events (SAEs) will be evaluated according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
  All adverse events occurring during the clinical trial will be recorded, including their clinical manifestations, severity, onset and resolution times, management measures, and outcomes. The correlation between AEs and the investigational drug will also be determined.

SECONDARY OUTCOMES:
Pharmacokinetic - Primary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  Cmax
Pharmacokinetic - Primary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  AUC(0-t)
Pharmacokinetic - Primary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  AUC(0-∞)
Pharmacokinetic - Secondary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  Tmax
Pharmacokinetic - Secondary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  AUC_%Extrap
Pharmacokinetic - Secondary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  CL
Pharmacokinetic - Secondary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  Vd
Pharmacokinetic - Secondary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  MRT
Pharmacokinetic - Secondary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  λz
Pharmacokinetic - Secondary Parameters | For healthy subjects: Predose and up to 24 hours postdose; For colorectal cancer subjects: Predose and up to 4 hours postdose
  T1/2

OTHER OUTCOMES:
Exploratory Endpoints | During Surgery
  Evaluation of Tumor Imaging Effects During Surgery
Exploratory Endpoints | Predose and up to 4 hours postdose
  Assessment of the Relationship Between SPN01 Plasma Concentration and QTc Interval Effects (if applicable)
Exploratory Endpoints | Predose and up to 4 hours postdose
  Qualitative and Quantitative Analysis of Metabolites from Blood/Urine Samples